CLINICAL TRIAL: NCT00769756
Title: Evaluation of Three New Strategies to Fight Obesity in Families
Status: Completed | Type: Observational
Sponsor: University of Magdeburg (Other)
Responsible Party: Prof. Dr. Claus Luley, MD, Institut of Clinical Chemistry, University Magdeburg
Other Study IDs: MD 22/06
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: Different Strategies to Fight Obesity in Families
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 2: Financial incentive
  For the parents the financial incentive was 5 euros for every kilogram of weight-loss. For children the weight loss was calculated differently, taking into account the individual need of each child to lose weight. Children with a body mass index between the 90th and 97th age-adjusted BMI-percentile were asked to maintain their weight, and were paid in dependence on how well they managed to achieve this goal. Children with age-adjusted BMI-percentiles between 97 and 99, or above the 99th age-adjusted BMI-percentile received 5 euros per weight losses of respectively 500 g or 1 kg.
- 1: The telemedical equipment consisted of a weighing scale for each family, an accelerometer for each participant, and a Homebox for each family which received the data from the scale and the accelerometers via bluetooth and transfered them via a telephone link to a server in Munich.
- 3: The basic diet for all participants was supported by a list giving the calorie contents of a large variety of food-stuffs. The dual diet group received a second list giving the glycemic index (GI) for a large variety of carbohy-drates. Emphasis was placed on a preference for low-GI carbohydrates but not on avoidance of carbohydrates as required by the Atkins diet.

SUMMARY:
Context: Endeavours to reduce overweight by calorie-restriction diets are often neither sufficient nor sustained. The growing obesity epidemic demands additional measures to enhance and sustain weight loss.

Objective: To evaluate three alternative weight-loss measures on top of a calorie-restriction diet.

Design, Setting, and Participants: Six-month randomized and controlled trial using a three-factorial design. The participants were 110 families with 142 obese parents and their 119 obese children.

DETAILED DESCRIPTION:
Intervention: All families kept to a calorie-restriction diet and were assigned at random to one or more of three additional weight-loss strategies: (1) a diet on top of calorie-restriction with preference for carbohydrates having a low glycemic index (dual diet), (2) financial incentive, and (3) continuous telemetric control of weight and physical activity (telemonitoring). The design made it possible to determine the effect of each single measure: financial incentive vs. no financial incentive (54 vs.56 families), calorie-restriction vs. dual diet (53 vs. 57 fami-lies) and telemonitoring vs. no telemonitoring (19 vs. 91 families). The design also allowed an assessment of the effects of combinations of the additional measures, each adapted for possible effects of the other factors.

Main Outcome In the parents the outcome variable at 6 months was the relative weight loss. In children, be-cause of their body growth, the outcome variable was the age-adjusted BMI standard deviation score (BMI-SDS). Analysis was done by three-factorial ANOVA and by a one-factorial ANOVA with the included Dunnett test as a post-hoc comparison, to distinguish between the effects of the different combinations of the additional strategies.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2

Exclusion Criteria:

* disease of kidney or liver

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The participating families were recruited by means of newspaper advertisements in the area around the German city of Magdeburg. The children had to be older than 7 years to ensure that they were able to read, and younger than 13 to minimize interferences due to puberty. 177 families responded by telephone and received a letter de-scribing the aim and character of the study. 110 families then decided to participate and were invited to the first of four meetings with intervals of one week between successive meetings.
Sampling Method: Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
In the parents the outcome variable at 6 months was the relative weight loss. In children, because of their body growth, the outcome variable was the age-adjusted BMI standard deviation score (BMI-SDS). | six and twelve month

SECONDARY OUTCOMES:
effects of the different combinations of the additional strategies to reduce weight | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Luley, MD, Principal Investigator — University Magdeburg, Germany
Locations (1):
- University Otto-von-Guericke, Magdeburg, Germany